CLINICAL TRIAL: NCT05187091
Title: The SWOAR Trial: A Phase III Trial Evaluating Sparing of Swallowing and Aspiration Related Organs at Risk & Submandibular Gland With Intensity Modulated Radiotherapy Versus Standard IMRT in Head and Neck Squamous Cell Carcinomas
Brief Title: The SWOAR Trial Sparing of Swallowing and Aspiration Related Organs at Risk & Submandibular Gland With Intensity Modulated Radiotherapy Versus Standard IMRT in Head and Neck Squamous Cell Carcinomas
Acronym: SWOAR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Aman Sharma, Assistant Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021/05/043810
Record Dates: First submitted 2021-08-18; First posted 2022-01-11 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Head and Neck Neoplasms; Swallowing Sparing IMRT
Keywords: IMRT; Dysphagia; Aspiration; Head and neck cancer; Radiation
MeSH Terms: conditions — Head and Neck Neoplasms; Deglutition Disorders | interventions — Deglutition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard IMRT (No Intervention): Standard IMRT with radical CRT/RT
- Swallowing Sparing IMRT (Experimental): Standard IMRT with radical CRT/RT with additional sparing of dysphagia-aspiration related structures & submandibular gland sparing by SWOAR-IMRT
  Interventions: Radiation: Swallowing and submandibular sparing IMRT

INTERVENTIONS:
Radiation: Swallowing and submandibular sparing IMRT — Standard IMRT with radical CRT/RT with additional sparing of dysphagia-aspiration related structures & submandibular gland sparing by SWOAR-IMRT
  Arms: Swallowing Sparing IMRT

SUMMARY:
The aim of SWOAR TRIAL is to test sparing of Dysphagia/ Aspiration risk structures (DARS) and contra lateral submandibular gland by IMRT. HNSCC of the oropharynx, larynx and the hypopharynx treated with radical concurrent chemoradiotherapy or radiotherapy will be included in the trial. Patients will be randomized to SWOAR IMRT or standard IMRT.

Swallowing function will be evaluated the MD Anderson Dysphagia Inventory (MDADI) scoring. Difference in the mean composite score of MDADI, a patient-reported outcome, at 6 months post radiotherapy is the primary outcome of the trial.

Secondary Objectives include longitudinal assessment of aspiration prevention as evaluated by FEES by the 8 point penetration-aspiration score. Swallowing function, will be assessed by using the MDADI at baseline, at completion of CRT/RT, 3, 6, 12, and 24 months.

Assessment of acute and late toxicity assessed at baseline, weekly during radiotherapy and then at 3, 6, 12, and 24 months post treatment as per RTOG and LENT SOMA score, respectively.

Treatment outcomes will be assessed in terms of loco-regional tumor recurrence and overall survival, assessed at follow-up visits 3, 6, 12, and 24 months post treatment and then annually until 5 years post treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 or above and less than 70 years
2. Patient undergoing radiotherapy for HNSCC of the Oropharynx or Larynx or Hypopharynx.
3. Stage T1-4, N0-3, M0 disease with histologically confirmed squamous cell carcinoma requiring bilateral neck radiotherapy and where sparing of contra lateral or one submandibular gland is possible
4. Radiotherapy with concomitant chemotherapy (unless contraindicated) is the planned treatment
5. Karnofsky performance score greater or equal 70
6. Available to attend long term follow- up;
7. Ability to complete the MD Anderson Dysphagia Inventory (MDADI) and EORTC quality of life questionnaires English or Hindi Version.
8. Willingness to undergo FEES.
9. Written informed consent for treatment.
10. Available to attend long term follow- up

Exclusion Criteria:

1. Early Carcinoma Glottis (T1-T2, N0M0)
2. Metastatic disease.
3. Previous radiotherapy to the head and neck region
4. Lateralised tumours, requiring unilateral irradiation
5. Patients requiring radiation to both submandibular glands
6. Evidence of pre-existing swallowing dysfunction (not related to HNC);
7. Major head and neck surgery (excluding biopsies/tonsillectomy);
8. Tracheostomy placement
9. Previous or concurrent illness, which in the investigator's opinion would interfere with completion of therapy, trial assessments or follow-up
10. Any invasive malignancy within previous 2 years (other than non melanomatous skin carcinoma or cervical carcinoma in situ).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2021-07-11 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change in swallowing function post radiotherapy | 6 months
  Primary objective of the SWOAR trial is to determine whether sparing the DARS by SWOAR IMRT, changes swallowing function compared to S- IMRT in advanced HNSCC. The impact of sparing the DARS with SWOAR-IMRT on late swallowing function will be evaluated the MDADI. Difference in the mean composite score of MDADI, a patient-reported outcome, at 6 months post radiotherapy is the primary outcome of the trial. MDADI score ranges from 0-100 where 0 is the worst and 100 is the best score for dysphagia assessment

SECONDARY OUTCOMES:
Swallowing assessment | longitudinal assessment till 2 years
  Swallowing will be assessed by using the MDADI at baseline, at completion of CRT/RT, 3, 6, 12, and 24 months.
Aspiration assessment | longitudinal assessment till 2 years
  Longitudinal assessment of aspiration prevention as evaluated by FEES by the 8 point penetration-aspiration score. Patients will be subjected to 10 ml of liquid, semi solid and solid meal at baseline, at completion of CRT/RT, 3, 6, 12 and 24 months.6, 12, and 24 months.
Acute Toxicity | longitudinal assessment till 2 years
  Assessment of acute weekly during radiotherapy as per RTOG
  RTOG grading is from 0 to IV where 0 represents no findings and IV being the worst Findings
Late Toxicity assessment by RTOG | longitudinal assessment till 2 years
  Assessment of late toxicity at 3, 6, 12, and 24 months post treatment as per RTOG score.
  RTOG is from 0 to IV where 0 represents no findings and IV being the worst Findings
Late Toxicity assessment by LENT SOMA | longitudinal assessment till 2 years
  Assessment of late toxicity at 3, 6, 12, and 24 months post treatment as LENT SOMA score.
  LENT SOMA score is from 0 to IV where 0 represents no findings and IV being the worst Findings
Treatment outcome: Loco-regional tumor control | 2 years
  Loco-regional tumor control at 2 years At follow up of 3, 6, 12, and 24 months post treatment
Treatment outcome: Overall survival | 2 years
  Overall survival at 2 years At follow up of 3, 6, 12, and 24 months post treatment
Quality of life assessment: EORTC QLQ C-30 | longitudinal assessment till 2 years
  EORTC QLQ C-30 questionnaire At follow up of 3, 6, 12, and 24 months post treatment The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items.
  Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. High score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Quality of life assessment: EORTC QLQ HN35 | longitudinal assessment till 2 years
  As per the EORTC QLQ HN35 questionnaire At follow up of 3, 6, 12, and 24 months post treatment The head & neck cancer module incorporates seven multi-item scales that assess pain, swallowing, senses (taste and smell), speech, social eating, social contact and sexuality. There are also eleven single items. For all items and scales, high scores indicate more problems (i.e. there are no function scales in which high scores would mean better functioning). The scoring approach for the QLQ-H&N35 is identical in principle to that for the symptom scales / single items of the QLQ-C30.

CONTACTS AND LOCATIONS:
Locations (1):
- Nci, Aiims, Jhajjar, Haryana, India

IPD SHARING:
Plan to Share IPD: No